CLINICAL TRIAL: NCT05495113
Title: In a Patient With Mild Dementia, Improvement of Cognitive Function Using YMS-201B, To Evaluate the Effectiveness and Safety, Randomized, Double-blinded, Sham Control Comparison, Confirmatory
Brief Title: The Efficacy and Safety of tDCS in Patients With Mild Dementia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ybrain Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YB_ST_SIT1901
Record Dates: First submitted 2022-01-19; First posted 2022-08-10 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Mild Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Stimulation (Sham Comparator): Sham Stimulation
  Interventions: Device: Sham stimulation using YMS-201B
- Real Stimulation (Active) (Experimental): transcranial Direct Current Stimulation (tDCS) application 5 ~7 days a week for 26 weeks
  Interventions: Device: YMS-201B (Device: Mind STIM)

INTERVENTIONS:
Device: YMS-201B (Device: Mind STIM) — transcranial Direct Current Stimulation (tDCS) 2mA for 30 min; 30 sec of ramp-up and -down; left (anode) and right (cathode) Dorsolateral prefrontal cortex (DLPFC)
  Arms: Real Stimulation (Active)
Device: Sham stimulation using YMS-201B — Sham stimulation; only 30 sec of ramp-up and -down; left (anode) and right (cathode) Dorsolateral prefrontal cortex (DLPFC)
  Arms: Sham Stimulation

SUMMARY:
This study evaluated the effectiveness and safety of improving Mild Dementia by applying tDCS for 26 weeks to patients with Mild Dementia.

DETAILED DESCRIPTION:
Patients received tDCS for 30 minutes with an intensity of 1.5 to 2 mA. tDCS was applied over the left (anode) and right (cathode) dorsolateral prefrontal cortex (DLPFC) 5~7 times a week and they were evaluated every 26weeks through questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 55 to 90 years old.
* Those diagnosed with dementia (major neurocognitive disorder, neurocognitive disorder) according to the criteria of Diagnostic and Statistical Manual (DSM-V) or The International Statistical Classification of Diseases and Related Health Provisions (ICD-10).
* Patients with mild dementia with a MMSE (Mini Mental State Examination) score of 18 points or more and less than 26 points) and less than 26 points.
* Person who has a clinical dementia rating (CDR) global score of 0.5 or 1.0, while CDR-SOB (Sum of Boxes) score satisfies 0.5 to 4.0 points 2)
* Acetylcholinease inhibitors (ACEI) and NMDA receptor inhibitors are those with the same usage and capacity for at least 3 months from the date of screening.

  * Patients who are taking drugs for cognitive functional treatment (e.g., pregabalin, gabapentincholinephocerate, etc.) other than acetylcholine inhibitor and NMDA receptor antagonist, and drugs for chronic diseases including hypertension, diabetes, hyperlipidemia, thyroid disease, etc.
* A person who can read and understand the subject's explanation and consent form, and who can speak at the level of ability to respond to questionnaires.
* A person who can be accompanied by a guardian when visiting a research institute during the clinical trial process, and who can help the guardian to proceed with the clinical trial process normally.
* A person who voluntarily decided to participate in this clinical trial and agreed in writing to the subject's written consent, who can participate in the pre-clinical trial period.

Exclusion Criteria:

* A person with a history of uniaxial psychiatric diseases including intellectual disability, schizophrenia, alcoholism, and bipolar disorder in the past.
* A person who has a history of convulsions within 5 years of screening.
* Those who have been diagnosed with severe cerebrovascular stenosis, subdural hemorrhage, brain tumor, and brain abscess through transient ischemic attack, stroke or MRI within one year from the screening date and are considered inappropriate for participation in this test.
* A person who has cerebral damage due to trauma, ischemia, hypoxia, etc.
* A person who has been hospitalized for mental or emotional problems within 5 years of screening.
* A person who abused drugs within 5 years of screening.
* A person who received treatment for alcoholism within 5 years of screening.
* A person who can't read even with glasses on due to poor eyesight.
* A person who can't understand a conversation because of hearing impairment even when wearing a hearing aid.
* A person who has difficulty breathing when sitting still.
* A person who attempted suicide within 6 months from the screening date.
* A person who is judged to have a problem with brain waves and direct current stimulation electrodes due to deformities, inflammatory reactions, or other dermatological problems in the scalp.
* A person who is judged to have other reasons for prohibition of use of tDCS medical devices (e.g., when a metal plate is inserted into the head, etc.).
* Those who participated in other clinical trials within 30 days of screening.
* Among female subjects who are likely to be pregnant, those who disagree with contraception* in a medically permitted manner during this clinical trial period.

  *Medically permitted contraceptive methods: condoms, oral contraceptives that last at least 3 months, injections or insertion contraceptives, etc. are used, and intrauterine contraceptives are installed, etc.
* Pregnant women or lactating women.
* In addition to the above, a person in charge of the test or a person in charge has a clinical significance that is medically judged and deemed inappropriate for this test.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in K-MMSE (Mini Mental State Examination) | After 26 weeks after treatment
  Changes in K-MMSE after 26 weeks form pretreatment (min value : 0 / max value: 30 / Higher scores mean a better outcome)

SECONDARY OUTCOMES:
Changes in K-IADL(Korean-Isturemental Activities of Daily Living) | After 26 weeks after treatment
  Changes in K-IADL after 26 weeks from pretreatment (min value : 0 / max value: 33 / Higher scores mean a worse outcome)
Changes in CDR(Clinical Dementia rating) | After 26 weeks after treatment
  Changes in CDR after 26 weeks from pretreatment (min value : 0 / max value: 3 / Higher scores mean a worse outcome)
Changes in MoCA-K (Korean version of Montreal Cognitive Assessment) | After 26 weeks after treatment
  Changes in MoCA-K after 26 weeks from pretreatment (min value : 0 / max value: 30 / Higher scores mean a better outcome)
Changes in NPI (Neuropsychiatric Inventory) | After 26 weeks after treatment
  Changes in NPI after 26 weeks from pretreatment (min value : 0 / max value: 144 / Higher scores mean a worse outcome)
Changes in QoL-AD(Quality of life-ADL-AD) | After 26 weeks after treatment
  Changes in QoL-AD after 26 weeks from pretreatment (min value : 13 / max value: 52 / Higher scores mean a better outcome)
Changes in FQoL-AD (Family's Quality of life-ADL-AD) | After 26 weeks after treatment
  Changes in FQoL-AD after 26 weeks from pretreatment (min value : 13 / max value: 52 / Higher scores mean a better outcome)
Changes in ADAS-Cog 11 (Alzheimer's Disease Assessment Scale-Cog 11) | After 26 weeks after treatment
  Changes in ADAS-Cog 11 after 26 weeks from pretreatment (min value : 0 / max value: 70 / Higher scores mean a worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: jung yong an, MD, Principal Investigator — Incheon St.Mary's Hospital
Locations (2):
- South Korea (2):
  - The Catholic University of Korea at incheon, Incheon
  - Korea University, Seoul

IPD SHARING:
Plan to Share IPD: No
to be determine